CLINICAL TRIAL: NCT04292821
Title: Performance Study of BIOPSY SCANNER LLTECH© Technology in the Immediate Diagnosis of Breast Cancer
Brief Title: BIOPSY SCANNER LLTECH© Technology for Diagnosis of Breast Cancer
Acronym: LLTECHBreast
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191059
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: breast lesion; breast cancer; B3 breast lesion; atypical breast lesion; breast imaging; one-day breast diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients consulting for breast lesion Bi Rads 4 or 5: Patients consulting for breast lesion Bi Rads 4 or 5

SUMMARY:
Breast cancer is a frequent pathology and the speed of initial diagnosis makes it possible to improve the course of care and to reduce the anxiety of the patients. For a complete assessment, several biopsies may be necessary, including lymph node biopsies. Once the histological sample has been taken, a preparation is necessary (time consuming technician) then a reading by a pathologist requiring at least 48-72h. Cytology allows immediate diagnosis, but it requires the presence of a pathologist in the collection room. Finally, some biopsies can be non-contributory (if there is not enough tissue removed) and require new samples. A tool allowing immediate control of the tissue and an initial diagnosis without mobilizing the pathologist (who will make the result complete with immunohistochemistry) would make it possible to anticipate the next course of care and facilitate treatment. The BIOPSY SCANNER LLTECH © technology would allow images on fresh unprepared tissue to obtain images allowing immediate diagnosis by a non-pathologist, the same tissue could then be technical for a complete analysis by the pathologist.

The investigators propose a study evaluating the diagnostic capacities by non pathologists from images obtained by the BIOPSY SCANNER LLTECH © technology on breast and lymph node biopsies. Based on this study, an atlas on breast lesions could be created to allow a broader evaluation of this technology in daily practice in diagnostic of breast pathology.

DETAILED DESCRIPTION:
In France, 59,000 new cases of breast cancer are diagnosed per year, but with systematic screening, more than 400,000 women will be biopsied each year. Less than 50% of women in France respond to organized screening and one of the reasons put forward is in particular the anxiety linked to waiting for the result of the biopsy if it turns out to be necessary.The BIOPSY SCANNER LLTECH © technology would allow images on fresh unprepared tissue to obtain images allowing immediate diagnosis by a non-pathologist (Annex 2: description of the manufacturer), the same tissue could then be technically analyzed for a complete analysis pathologic.

The BIOPSY SCANNER LLTECH © is an optical imaging device for the microscopic evaluation of deep tissue samples. It enables rapid imaging of samples on a cellular scale, in a non-invasive and non-destructive manner, and to reveal their microarchitecture and cellular organization.

The Biopsy Scanner uses the patented technique of full field white light interferometry. This technique is considered to be the equivalent of optical resolution ultrasound (≈ 1 μm) in 3 directions. A sample placed in the system is illuminated by an inconsistent light source.

The light reflected by the sample is collected by the interferometer and interferes with the light reflected by a reference mirror. This interference signal is recorded by a camera. The interferometric technique and the coherence properties of the light source make it possible to select the signal which comes from a limited volume in the depth of the sample. This property of the system is called optical sectioning and ensures good axial imaging resolution (1 μm). The transverse resolution is good (1.5 μm) thanks to the integration of microscope objectives in the interferometer.

Currently, it is necessary for an immediate diagnosis of breast cancer to have a second expert cytologist doctor (it is a difficult learning technique) in the radiologist's room to check that the tissue removed is sufficient. In addition, a second sample is necessary to obtain a complete histology. The BIOPSY SCANNER LLTECH © technology could allow patients to be informed more quickly while avoiding mobilizing on-site expertise and taking 2 samples.The investigators hypothesize that the BIOPSY SCANNER LLTECH © technique will allow the radiologist to provide immediately after the breast or lymph node biopsy, on fresh unprepared tissue, a positive or negative diagnosis of cancer, with sufficient diagnostic performance to consider its generalization.

The study will also allow us to see whether a learning curve is necessary and to assess its duration. It should be noted that there is no reason to think a priori that the sensitivities / specificities will be different depending on the type of biopsy (breast or lymph node) which will therefore be analyzed in the same group in the main analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old requiring a breast biopsy for an birads 4 or 5 nodular radiological lesion or lymph node for a lymph node judged to be radiologically suspect (cortex thickened by more than 3 mm)

Exclusion Criteria:

* Patients under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients consulting for breast lesion Bi Rads 4 or 5
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value (PPV) | At the end of inclusion time
  Positive predictive value (PPV) of the diagnosis of breast cancer by the analysis of images BIOPSY SCANNER LLTECH © carried out by a senior radiologist taking as reference the results provided by histology on tissue section.

SECONDARY OUTCOMES:
Reproductibility | At the end of inclusion time
  Comparison of sensitivity, specificity, positive predictive value and negative predictive value of the diagnosis of breast cancer by the analysis of BIOPSY SCANNER LLTECH © images by a junior radiologist versus senior radiologist versus pathologist versus surgeon
Efficiency for each histologic type | At the end of inclusion time
  Comparison of sensitivity, specificity, positive predictive value and negative predictive value of the diagnosis of breast cancer by the analysis of BIOPSY SCANNER LLTECH © images according to the histological characteristics of the tumor (according to grade, according to luminal A / luminal B profile / triple negative / HEr2 3+)
Efficiency compared between breast tissue and lymph node | At the end of inclusion time
  Comparison of the sensitivity, specificity, positive predictive value and negative predictive value of the diagnosis of breast cancer by the analysis of BIOPSY
Progression curve | At the end of inclusion time
  Number of samples required to reach the objective of the same diagnostic capacity as the pathologist from these images
Image atlas | At the end of inclusion time
  Establishment of an image atlas facilitating the subsequent use of this technology by non-pathologists
Image recognition algorithm | At the end of inclusion time
  Implementation of an image recognition algorithm for automated diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Catherine UZAN, Md PhD, Principal Investigator — Pitié-Salpêtrière Hospital (AP-HP)
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Simon A, Badachi Y, Ropers J, Laurent I, Dong L, Da Maia E, Bourcier A, Canlorbe G, Uzan C. Value of high-resolution full-field optical coherence tomography and dynamic cell imaging for one-stop rapid diagnosis breast clinic. Cancer Med. 2023 Oct;12(19):19500-19511. doi: 10.1002/cam4.6560. Epub 2023 Sep 29. PMID 37772663